CLINICAL TRIAL: NCT03351036
Title: Evaluation of the S3 Guideline on Avoidance of Perioperative Hypothermia - Already a Standard or Wishful Thinking?
Status: Withdrawn | Type: Observational
Why Stopped: Change in personnel
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Timo Iden, Dr. med., University Hospital Schleswig-Holstein
Other Study IDs: S3_Evaluation_Hypothermia
Record Dates: First submitted 2015-12-07; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Hypothermia; Perioperative/Postoperative Complications; Hypothermia Following Anesthesia
Keywords: Hypothermia
MeSH Terms: conditions — Hypothermia; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Perioperative hypothermia is a common problem in today´s surgical and anesthesiological patient care and is associated with many adverse events. The intention of this study was to evaluate the current S3 guideline on the avoidance of perioperative hypothermia concerning it´s implementation in the clinical routine.

DETAILED DESCRIPTION:
Perioperative hypothermia is a common problem in today´s surgical and anesthesiological patient care and is associated with many adverse events such as impaired coagulation, increased risk for wound infections and patient discomfort among others. The intention of this study was to evaluate the current S3 guideline on the avoidance of perioperative hypothermia published in 2014 concerning it´s implementation in the clinical routine. In a first phase the current status should be recorded. If this reveals an inappropriate high incidence of perioperative hypothermia training arrangements shall be taken for non-physician personnel in the PACU in a 2nd phase of the project. The third phase is intended to evaluate the effect of the training arrangements on the incidence of hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years undergoing elective surgery admitted to the PACU

Exclusion Criteria:

* Patients < 18 years
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients ≥ 18 years undergoing elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative hypothermia | Immediately after arrival at PACU
  Evaluation of the S3 guideline on avoidance of perioperative hypothermia

SECONDARY OUTCOMES:
Incidence of intraoperative hypothermia | Duration of surgical procedure
  Evaluation of the S3 guideline on avoidance of perioperative hypothermia
Incidence of preoperative hypothermia | Immediately after arrival at holding area
  Evaluation of the S3 guideline on avoidance of perioperative hypothermia

CONTACTS AND LOCATIONS:
Overall Officials: Jan Höcker, MD, Study Director — Klinik für Anästhesiologie und Operative Intensivmedizin, Arnold-Heller-Str. 3, Haus 12, 24105 Kiel
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Torossian A, Brauer A, Hocker J, Bein B, Wulf H, Horn EP. Preventing inadvertent perioperative hypothermia. Dtsch Arztebl Int. 2015 Mar 6;112(10):166-72. doi: 10.3238/arztebl.2015.0166. PMID 25837741
- See also: S3 guideline (German) — http://www.awmf.org/leitlinien/detail/ll/001-018.html